CLINICAL TRIAL: NCT00348283
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab Endoscopy Trial to Evaluate the Effects on Mucosal Healing in Subjects With Crohn's Disease Involving the Colon
Brief Title: Effects of Adalimumab on Mucosal Healing in Subjects With Crohn's Disease Involving the Colon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Roopal B. Thakkar, M.D., Project Director Humira Gastroenterology, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-769
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double Blind (Placebo Comparator): Blinded study through Week 52. Adalimumab compared to placebo during blinded portion.
  Interventions: Biological: adalimumab; Biological: placebo
- Open Label (Other): Note: No comparator was used in Open-Label portion of study. From Week 8, subjects could have switched to open-label (OL) adalimumab 40mg administered subcutaneously (SC) every other week (eow)or OL adalimumab 40 mg SC every week (ew) dosing to treat disease flare or non-response. At Week 52, all remaining subjects were allowed to switch to the Open-Label portion of the study.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — At Baseline (Week 0), subjects received an OL dose of 160 mg adalimumab SC followed by an OL dose of 80 mg adalimumab SC at Week 2 (induction dose). At Week 4, subjects were randomized to either adalimumab 40 mg SC eow or placebo SC eow. Adalimumab 40 mg eow dosing through blinded portion of study, which continued through Week 52. While all subjects began blinded study drug (placebo or adalimumab), subjects could have switched to an OL dose of adalimumab upon disease flare or non-response at or after Week 8.
  Other Names: ABT-D2E7; Humira
  Arms: Double Blind
Biological: placebo — At Baseline (Week 0), subjects received an OL dose of 160 mg adalimumab SC followed by an OL dose of 80 mg adalimumab SC at Week 2 (induction dose). At Week 4, subjects were randomized to either adalimumab 40 mg SC eow or placebo SC eow. Placebo SC eow dosing through blinded portion of study, which continued through Week 52. While all subjects began blinded study drug (placebo or adalimumab), subjects could have switched to an OL dose of adalimumab upon disease flare or non-response at or after Week 8.
  Arms: Double Blind
Biological: adalimumab — At Baseline (Week 0), subjects received an OL dose of 160 mg adalimumab SC followed by an OL dose of 80 mg adalimumab SC at Week 2 (induction dose). At Week 4, subjects were randomized to either adalimumab 40 mg SC eow or placebo SC eow. Adalimumab or placebo SC eow dosing through blinded portion of study, which continued through Week 52. While all subjects began blinded study drug (placebo or adalimumab), subjects could have switched to an OL dose of adalimumab upon disease flare or non-response at or after Week 8. In the Open-Label arm, interventions were either adalimumab 40 mg SC eow or adalimumab 40 mg SC weekly. There was no placebo intervention post Week 52.
  Other Names: ABT-D2E7; Humira
  Arms: Open Label

SUMMARY:
The goal of this study was to test whether adalimumab can induce mucosal healing in subjects with moderate to severe ileocolonic Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease for greater than 4 months.
* A diagnosis of ileocolonic Crohn's Disease confirmed by endoscopy or radiologic evaluation within 3 years of Baseline.
* For subjects who have had operations in the ileocolonic region of the intestine after documented diagnosis of ileocolonic disease, postoperative recurrence of the disease must be documented.
* Endoscopic documentation of ulceration at Screening corresponding to a score of 2 or 3 in at least one of the five segments of the colon on the Ulcerated Surface subscore of the Simple Endoscopic Score for Crohn's Disease (SES-CD).
* Crohn's Disease Activity Index (CDAI) score of >= 220 and <= 450.
* Males and females >= 18 and <= 75 years of age at the Baseline visit.
* Adequate cardiac, renal and hepatic function as determined by the Principal Investigator and demonstrated by Screening laboratory evaluations, questionnaires, and physical examination results that do not indicate an abnormal clinical condition which would place the subject at undue risk and thus preclude subject participation in the study.
* Subjects must be able to self-inject study medication or have a designee or healthcare professional who can inject the study medication.
* Subjects must agree to undergo up to 4 endoscopies.

Exclusion Criteria:

* History of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinoma - in-situ of the cervix.
* History of listeria, human immunodeficiency virus (HIV), hepatitis B, an immunodeficiency syndrome, central nervous system (CNS) demyelinating disease, or untreated tuberculosis (TB).
* Subject with a current diagnosis of ulcerative colitis or indeterminate colitis as determined by the Investigator and Abbott Medical Monitor.
* Subject who has had surgical bowel resections within the past 6 months or is planning any resection at any time point while enrolled in the study.
* Subject with an ostomy or ileoanal pouch. (Subjects with a previous ileo-rectal anastomosis are not excluded).
* Subject who has received any investigational biological agent in the past 3 months or 5 half-lives prior to Baseline (whichever is longer).
* Subjects with a poorly controlled medical condition and any other condition which, in the opinion of the Investigator or the sponsor, would put the subject at risk by participation in the protocol.
* Subject who has previously used infliximab or any anti-TNF (anti tumor necrosis factor), even investigational, within 8 weeks of Baseline.
* Subject who has previously used infliximab or any anti-TNF agent and has not clinically responded.
* Previous treatment with adalimumab or previous participation in an adalimumab clinical study.
* Subjects on prednisone > 40 mg/day (or equivalent).
* Subjects on budesonide > 9 mg/day.
* Subjects with any prior exposure to Tysabri® (natalizumab).
* Subjects with a previous history of dysplasia of the gastrointestinal tract, or found to have dysplasia in any biopsy performed during the Screening endoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Andrée Camez, Study Director — Abbott
Locations (21):
- United States (7):
  - Atlanta, Georgia
  - Chicago, Illinois
  - Chevy Chase, Maryland
  - Plymouth, Minnesota
  - Rochester, Minnesota
  - Mexico, Missouri
  - Great Neck, New York
- Vienna, Austria
- Belgium (3):
  - Bonheiden
  - Leuven
  - Roeselare
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
- Lille, France
- Germany (3):
  - Berlin
  - Hamburg
  - Kiel
- Torino, Italy
- Amsterdam, Netherlands

REFERENCES:
- [Derived] Sandborn WJ, Lewis JD, Panes J, Loftus EV, D'Haens G, Yu Z, Huang B, Lacerda AP, Pangan AL, Feagan BG. Association Between Proposed Definitions of Clinical Remission/Response and Well-Being in Patients With Crohn's Disease. J Crohns Colitis. 2022 Mar 14;16(3):444-451. doi: 10.1093/ecco-jcc/jjab161. PMID 34546360
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Rutgeerts P, Reinisch W, Colombel JF, Sandborn WJ, D'Haens G, Petersson J, Zhou Q, Iezzi A, Thakkar RB. Agreement of site and central readings of ileocolonoscopic scores in Crohn's disease: comparison using data from the EXTEND trial. Gastrointest Endosc. 2016 Jan;83(1):188-97.e1-3. doi: 10.1016/j.gie.2015.06.018. Epub 2015 Jul 30. PMID 26234693
- [Derived] Colombel JF, Rutgeerts PJ, Sandborn WJ, Yang M, Camez A, Pollack PF, Thakkar RB, Robinson AM, Chen N, Mulani PM, Chao J. Adalimumab induces deep remission in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2014 Mar;12(3):414-22.e5. doi: 10.1016/j.cgh.2013.06.019. Epub 2013 Jul 12. PMID 23856361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were to be enrolled in 9 countries. Subjects were enrolled at 19 sites in 8 countries. No subjects were enrolled in Sweden.
Pre-assignment Details: All subjects (135 subjects) enrolled in the study received an open-label dose of 160 mg adalimumab subcutaneously (SC) at Baseline (Week 0) followed by 80 mg adalimumab SC at Week 2 (induction dose). At Week 4, subjects were randomized to either adalimumab 40 mg SC every other week (eow) or placebo SC eow(129 subjects).
Groups:
- Placebo: SC dosing eow
- Adalimumab: 40 mg SC eow
Period: Induction
Arm/Group | Placebo | Adalimumab
Started | 0 | 135 (Subjects received an open- label dose of 80 mg adalimumab at Week 2 (induction dose).)
Completed | 0 | 129 (Subjects provided more than one reason for discontinuing during induction.)
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 4
Period: Double Blind
Arm/Group | Placebo | Adalimumab
Started | 65 (At Week 4, subjects were randomized to either adalimumab 40 mg eow or placebo eow.) | 64 (At Week 4, subjects were randomized to either adalimumab 40 mg eow or placebo eow.)
Completed | 60 | 54
Not Completed | 5 | 10
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Pregnancy | 0 | 1
Period: Open Label
Arm/Group | Placebo | Adalimumab
Started | 0 (No comparator was used in the Open Label portion of the study.) | 100 (14 subjects completed the Double Blind portion of the study but did not enter the Open Label period.)
Completed | 0 | 66
Not Completed | 0 | 34
Not completed — Adverse Event | 0 | 8
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 13
Not completed — Administrative reasons | 0 | 5
Not completed — Subject moved to the United States | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Sponsor decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo; Adalimumab 40 mg Every Other Week: At Baseline (Week 0), subjects received an OL dose of 160 mg adalimumab SC followed by an OL dose of 80 mg adalimumab SC at Week 2 (induction dose). At Week 4, subjects were randomized to either adalimumab 40 mg SC eow or placebo SC eow.
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab 40 mg Every Other Week | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 63 | 62 | 125
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 37.2 (12.60) | 37.1 (11.10) | 37.1 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 6
  United States | 20 | 12 | 32
  Canada | 22 | 18 | 40
  Belgium | 14 | 25 | 39
  Austria | 2 | 0 | 2
  Netherlands | 1 | 2 | 3
  Germany | 1 | 1 | 2
  Italy | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Without Mucosal Ulceration at Week 12
Description: Subjects were to have undergone up to 4 endoscopies to evaluate the presence or absence of mucosal ulceration: at Screening, at Week 12 (subjects who moved to open label (OL) drug between Week 8 and Week 12 because of disease flare or non-response were evaluated by endoscopy prior to receiving OL dosing), at the time of switch from blinded study drug to OL adalimumab at any time after Week 12, and at Week 52 or Early Termination. Subjects who remained blinded for the entire 52-week trial or switched to OL adalimumab between Week 8 and Week 12 were to have undergone 3 endoscopies.
Time Frame: Week 12
Population: Analysis was on ITT subjects with mucosal ulceration at Screening. Subjects who did not have endoscopy at Week 12 were considered to have mucosal ulceration at Week 12 (NRI). If subjects had endoscopy at Week 8, the endoscopy results from Week 8 were carried forward to Week 12 for the primary efficacy analysis.
Measure: Number; unit: Subjects
Groups:
- Adalimumab: 40 mg every other week
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 61 | 62
Subjects | 8 | 17
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; ITT population: all subjects randomized at Week 4 who had at least 1 dose of blinded therapy. The sample-size (placebo = 65 subjects; adalimumab = 65 subjects) for the primary efficacy analysis was calculated using 88% power at 0.05 alpha level based on the assumption that 25% and 5% of subjects were without mucosal ulceration at Week 12 in adalimumab 40 mg eow and placebo groups, respectively. However, subjects without mucosal ulceration at Screening were excluded from the primary analysis; Test type: Superiority or Other; p = 0.056, Cochran-Mantel-Haenszel — The P value is from Cochran-Mantel-Haenszel test with clinical response (CR-70 responder status) at Week 4 as the stratification factor; Because of the hierarchical testing scheme used for testing the ranked secondary endpoints, alpha level of 0.05 was used at each stage of testing

2. Secondary Outcome: Number of Subjects With Clinical Remission Crohn's Disease Activity Index (CDAI) < 150 at Week 12
Description: Clinical remission is defined as a CDAI less than 150. A lower score correlates with less severe Crohn's disease activity. The CDAI range for this study was 0 to 961.
Time Frame: Week 12
Population: ITT set. NRI method was used to impute the missing values.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 65 | 64
Subjects | 18 | 30
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; The null hypothesis was that there is no difference in proportion of subjects with clinical remission at Week 12 in the two treatment groups; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects Without Mucosal Ulceration at Week 52
Description: The number of subjects receiving blinded study drug in each treatment group who were without mucosal ulceration at Week 52.
Time Frame: Week 52
Population: The secondary efficacy analysis included the ITT subjects who had mucosal ulceration at screening. NRI method was used to impute the missing values.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 61 | 62
Subjects | 0 | 15
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; The null hypothesis was that there is no difference between proportions of subjects without mucosal ulceration at Week 52 in the two treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Subjects With Clinical Remission (CDAI < 150) at Week 52
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) less than 150. A lower score correlates with less severe Crohn's disease activity. The CDAI range for this study was 0 to 961.
Time Frame: Week 52
Population: ITT set. NRI method was used to impute the missing values.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 65 | 64
Subjects | 6 | 21
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; The null hypothesis was that there is no difference in proportion of subjects with clinical remission at Week 52 in the two treatment groups; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Subjects Without Mucosal Ulceration at Both Week 12 and Week 52
Description: The number of subjects receiving blinded study drug in each treatment group who were without mucosal ulceration at both Week 12 and Week 52.
Time Frame: Weeks 12 and 52
Population: Analysis was on ITT subjects who completed the Double Blind period and had Week 52 evaluations while in the Double Blind period. NRI method was used to impute the missing values.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 11 | 25
Subjects | 0 | 7
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; The null hypothesis was that there is no difference between proportions of subjects without mucosal ulceration at both Week 12 and Week 52 in the two treatment groups; Test type: Superiority or Other; p = 0.150, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Subjects With Clinical Remission (CDAI < 150) at Both Week 12 and Week 52
Description: as for outcome 4
Time Frame: Weeks 12 and 52
Population: ITT set. NRI method was used to impute the missing values.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 65 | 64
Subjects | 3 | 19
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Serious adverse events were not assessed for placebo subjects (Total at risk = 0) as all subjects received an OL dose of 160 mg adalimumab at Week 0 followed by an OL induction dose of 80 mg adalimumab at Week 2.
Groups:
- Adalimumab: All subjects (135 subjects) enrolled in the study received adalimumab 160 mg at Baseline followed by adalimumab 80 mg at Week 2 (Induction dose).
Arm/Group | Placebo | Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/0 | 20/135
Other Adverse Events (participants affected / at risk) | 43/65 | 49/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=0) | Adalimumab (N=135)
Coronary artery disease (Cardiac disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 8
Ileal stenosis (Gastrointestinal disorders) | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Clostridium difficile toxin test positive (Investigations) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Adalimumab (N=64)
Abdominal distension (Gastrointestinal disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Constipation (Gastrointestinal disorders) | 0 | 4
Crohn's disease (Gastrointestinal disorders) | 19 | 15
Flatulence (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 2 | 7
Influenza like illness (General disorders) | 3 | 6
Pyrexia (General disorders) | 4 | 2
Gastroenteritis (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 8 | 9
Sinusitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Headache (Nervous system disorders) | 6 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide ABBOTT at least sixty (60) days prior to submission for review, ABBOTT shall return within sixty (60) days. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period